CLINICAL TRIAL: NCT04625946
Title: Metformin as an Adjunctive Therapy to Catheter Ablation in Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hakan Oral, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00174848
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
Keywords: ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Standard of care ablation with recommendations for lifestyle modification and metformin.
  Interventions: Drug: Metformin; Behavioral: Recommendations for lifestyle modification.; Device: AliveCor
- Standard of care (Other): Standard of care ablation with recommendations for lifestyle modification.
  Interventions: Behavioral: Recommendations for lifestyle modification.; Device: AliveCor

INTERVENTIONS:
Drug: Metformin — Metformin immediate release will be initiated at 250 milligrams (mg) daily (orally), and increased as tolerated to 2000 mg daily over a four week period. If a patient is unable to tolerate a dose increase they will return to their last tolerated dose after omitting one days dosing. 0 to Six weeks after the initiation of drug the patient will undergo (standard of care) ablation with the intent of achieving rhythm control.
  Participants will stay on the metformin 12 months after the ablation. In addition, all participants will receive education on lifestyle changes and exercise which are standard of care as well as have a discussion with their treating electrophysiologist and receive a handout.
  Other Names: Glucophage
  Arms: Metformin
Behavioral: Recommendations for lifestyle modification. — All subjects will receive education on lifestyle changes and exercise which are standard of care. This will include discussion with their treating electrophysiologist and a handout.
Device: AliveCor — Device will be used in order to record an electrocardiogram during symptoms perceived to be AF. All patients will be instructed to transmit at least once per week.

SUMMARY:
This clinical trial is being done to determine if metformin, a drug which is normally used in diabetes, can reduce atrial fibrillation in patients who are having an ablation for atrial fibrillation (AF). Atrial fibrillation is an abnormal heart rhythm which research has shown is related in part to obesity and diabetes.

It is anticipated that the participants treated in the metformin arm will have greater freedom from recurrent atrial arrhythmias after ablation.

Eligible participants enrolled in the trial will be assigned to one of the treatment arms (no treatment or metformin) and have follow-up visits up to approximately 1 year after the ablation. Additionally, all patients will also receive education on lifestyle changes and exercise which are standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) >25 kilograms / square meter (kg/m2) with plan for rhythm control of atrial fibrillation by catheter ablation
* All subjects must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Individuals who are already taking metformin or other antidiabetic medications, including insulin
* Known diabetes
* Known allergy or Food and Drug Administration (FDA)-labeled contraindication to taking metformin (estimated glomerular filtration rate (eGFR)<30 millilitres per minute (mL/min)/1.73 square meters (m2), hypersensitivity to metformin, acute or chronic metabolic acidosis)
* Patients taking carbonic anhydrase inhibitors
* eGFR below 30 mL/min per 1.73 m2 or other clinical diagnosis of advanced renal disease
* Acute or chronic metabolic acidosis (serum bicarbonate <22 milliequivalents per liter (mEq/L))
* History of significant alcohol use (>2 drinks/day on average)
* History of hepatic dysfunction (serum bilirubin 1.5 times greater than ULN)
* History of New York Heart Association (NYHA) Class III or IV heart failure
* Pregnancy or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Freedom from recurrent atrial arrhythmias by 12 months after a single ablation to eliminate AF | 12 months after ablation
  There will be a 3 month blanking period after ablation during which recurrent atrial arrhythmias will not contribute to the primary endpoint.

SECONDARY OUTCOMES:
Time to recurrence of atrial fibrillation after a 3 month blanking period of ablation | up to 1 year after after ablation
Freedom from recurrent atrial arrhythmias at 1 year after ablation after the blanking period of 3 months | 6 months after ablation
Freedom from recurrent atrial arrhythmias at 6 months after repeat ablation | 6 months after a repeated ablation
Atrial Fibrillation Severity Score (AFSS) | up to 12 months after ablation
  There are a total of 19 questions (parts A,B, and C) in this questionnaire. This collects information regarding the participants atrial fibrillation. It includes seven questions for subjects to report severity of symptoms (i.e. palpitations, shortness of breath at rest/physical activity, exercise intolerance, fatigue at rest, and lightheadedness/dizziness, chest pain or pressure) on a Likert scale from 0 (subject did not have this symptom) to 5 (symptom bothers subject a great deal).
Percent change in weight at 3 months after ablation | 3 months after ablation
Percent change in weight at 6 months after ablation | 6 months after ablation
Percent change in hemoglobin A1c at 6 months after ablation | 6 months after ablation
Percent change in hemoglobin A1C at 12 months after ablation | 12 months after ablation
Incidence of major procedural complications | up to 30 days
  Complications include but are not limited to major bleeding, vascular injury, myocardial perforation, stroke, and mortality.
Atrial Fibrillation related morbidity during follow-up | up to approximately 1 year after ablation
  During follow-up visits information will be collected regarding Emergency department visits and hospital admissions due to AF, Transient Ischemic Attack (TIA)/cerebrovascular accident (CVA), and mortality. These will be collected as total numbers between groups.
Burden of Atrial Fibrillation assessed by AliveCOR Kardia Devices | 6 months after ablation
Burden of Atrial Fibrillation assessed by AliveCOR Kardia Devices | 1 year after ablation
Burden of Atrial Fibrillation assessed by AliveCOR Kardia Devices | 3 months after ablation

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Oral, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No